CLINICAL TRIAL: NCT05314504
Title: A Multicenter, Randomized, Rater-Blinded, No-Treatment Control Design Clinical Investigation to Evaluate the Effectiveness and Safety of YVOIRE Y-Solution 360 for Lip Augmentation
Brief Title: Clinical Investigation of YVOIRE Y-Solution 360 for Lip Augmentation in China
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: LG Chem (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: LG-HACL031
Record Dates: First submitted 2022-03-30; First posted 2022-04-06 (Actual); Last update posted 2024-12-19 (Actual); Status verified 2024-12

CONDITIONS: Lip Augmentation

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Test group (Experimental): Treatment administration to subjects
  Interventions: Device: YVOIRE Y-Solution 360
- Control group (No Intervention): After primary endpoint evaluation, eligible subjects will receive treatment at Week 12

INTERVENTIONS:
Device: YVOIRE Y-Solution 360 — Cross-linked sodium hyaluronate gel for injection with lidocaine
  Arms: Test group

SUMMARY:
To evaluate the effectiveness and safety of the investigational medical device, injected into the lips.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female adults 18 to 65 years of age (inclusive).
2. Subjects whose volume of the overall lips corresponds to score of 0 (none/minimal), 1 (mild), 2 (moderate), or 3 (pronounced) of the 5-point LFRS as assessed by the blinded Evaluating Investigator at Visit 1 (Screening).
3. Subjects who want a filler injection procedure for at least a 1-grade increase on the overall LFRS score after treatment.
4. Subjects who are informed of the purpose, method, and effectiveness of the clinical investigation and who sign the written informed consent form (ICF).
5. Except for surgically sterile male or female subjects, and female subjects with natural menopause (without drug intervention) for more than 2 years after last menstruation, other male or female subjects must agree to use an effective method throughout the entire clinical investigation period to prevent pregnancy

Exclusion Criteria:

1. Subjects who have lip tattoos, piercings, facial hair, or scars that would interfere with visualization of the lips and perioral area.
2. Subjects who have dentures or any device covering all or part of the upper palate, and/or severe malocclusion or dentofacial or maxillofacial deformities.
3. Subjects who have undergone oral surgery (e.g., tooth extraction, orthodontia, or implantation) within 6 months before enrollment or is planning to undergo any of these procedures during the clinical investigation.
4. Subjects who have received permanent facial implants or fillers (e.g., polymethylmethacrylate, silicone, polytetrafluoroethylene, autologous fat) in the face or neck, or are planning to be implanted with any of these products during the clinical investigation.
5. Subjects who have received non-permanent filler treatment in the lower face (below the orbital rim) or are planning to undergo during the clinical investigation, including but not limited to receiving calcium hydroxylapatite or poly-L lactic acid within 24 months before enrollment, or hyaluronic acid [HA] or collagen within 12 months before enrollment.
6. Subjects who have undergone the following procedure within 6 months before enrollment or are planning to undergo during the clinical investigation: Facial tissue augmentation or facial treatment with fat or botulinum injections in the lower face (below the orbital rim). messotherapy, face lift, stripping laser, dermabrasion, moderate or greater depth chemical peel, or other ablative procedures in face or neck.
7. Subjects who have used non-implantable lip plumping products within 10 days before enrollment anywhere in the treatment area or are planning to receive such treatment/intervention during the clinical investigation participation.
8. Subjects who have used any over-the-counter or prescription, oral or topical anti-wrinkle products for the lips or around the mouth within 3 months before enrollment or are planning to use such products during the clinical investigation.
9. Subjects who are on an ongoing regimen of anti-coagulation therapy (e.g., warfarin) or non-steroidal anti-inflammatory drugs (NSAIDs; e.g., aspirin, ibuprofen) or other substances known to increase coagulation time (e.g., herbal supplements with gingko biloba) within 10 days of undergoing investigational medical device injections.
10. Subjects who have history of anaphylaxis, multiple several allergies, or allergy to lidocaine, or amide local anesthetics, HA products, or Streptococcal protein, or are planning to undergo desensitization therapy during the clinical investigation.
11. Subjects with active inflammation, infection sites or unhealed wound in the mouth area.
12. Subjects who have history of herpetic eruption.
13. Subjects who have history of bleeding disorder based on the coagulation laboratory test results (international normalized ratio [INR], prothrombin time, and activated partial thromboplastin time [aPTT]) as per Investigator's discretion.
14. Subjects with abnormal laboratory assessment and judged clinically significant per Investigator's discretion (e.g., alanine aminotransferase [ALT] ≥ 2.5×upper limit of normal [ULN], aspartate aminotransferase [AST] ≥ 2.5×ULN).
15. Subjects who have porphyria.
16. Subjects who have a tendency to develop hypertrophic scar or keloid.
17. Subjects who have severe cardiovascular, hepatic or renal diseases considered as per Investigator's discretion.
18. Subjects who have malignant tumors or cancerous or precancerous lesion which could affect the clinical investigation.
19. Subjects who have untreated epilepsy.
20. Subjects who are ineligible for this clinical investigation as per Investigator's discretion.
21. Subjects who have participated in another clinical investigation within 1 month prior to Visit 1 (Screening).

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 174 (Actual)
Dates: Start 2022-01-11 (Actual); Primary Completion 2023-02-23 (Actual); Study Completion 2024-02-21 (Actual)

PRIMARY OUTCOMES:
Overall LFRS responder rate | at 12 weeks
  at 12 weeks after the last injection for the test group and at Week 12 for the control group

CONTACTS AND LOCATIONS:
Locations (1):
- Huashan Hospital Affiliated to Fudan University, Shanghai, China

IPD SHARING:
Plan to Share IPD: No